CLINICAL TRIAL: NCT06855745
Title: A Phase 2, Randomized, Double-blind, Multicenter Study to Assess the Safety and Efficacy of Topical Zabalafin Hydrogel Versus Vehicle in the Treatment of Participants With Mild to Moderate Atopic Dermatitis (CLEAR-AD1)
Brief Title: Phase 2 Randomized Double-blind Study to Assess Topical Zabalafin Hydrogel Vs Vehicle in Mild to Moderate AD.
Acronym: CLEAR-AD1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alphyn Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-101-003-00
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis (Eczema); Atopic Dermatitis Eczema; Atopic Dermatitis; Atopic Dermatitis (AD); Eczema; Eczema, Atopic
Keywords: Eczema; Childhood eczema; Adult eczema; AD; Dermatitis; Infected dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis

STUDY DESIGN:
Intervention Model Description: This is a randomised, double blind study aiming to enrol 72 participants across 10 sites in Australia. There are 2 cohorts: Cohort 1: Mild to moderate atopic dermatitis Cohort 2: Mild to moderate atopic dermatitis - with secondary skin infection. Once assigned to a cohort participants will be randomised into 1 of 2 Groups: Arm A: Zabalafin hydrogel or Arm B: vehicle (placebo). Randomisation will be 2:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Zabalafin 9.5%
  Interventions: Drug: zabalafin
- Arm B (Placebo Comparator): Placebo (vehicle)
  Interventions: Drug: zabalafin

INTERVENTIONS:
Drug: zabalafin — Active IP
  Other Names: AB-101

SUMMARY:
A Phase 2b study investigating the efficacy of zabalafin in people with mild to moderate atopic dermatitis (eczema).

DETAILED DESCRIPTION:
This is a randomised, double blind study aiming to enroll 72 participants across 10 sites in Australia. There are 2 cohorts: Cohort 1: Mild to moderate atopic dermatitis Cohort 2: Mild to moderate atopic dermatitis - with secondary skin infection. Once assigned to a cohort participants will be randomised into 1 of 2 Groups: Arm A: Zabalafin hydrogel or Arm B: vehicle (placebo). Randomisation will be 2:1 ratio. There is up to 2 weeks for screening and study treatment period of 16 weeks. Participants will need to attend the site every 2 weeks for 1 month and then monthly until Week 16 (end of study treatment). The primary objective (efficacy) will be assessed using validated Investigators Global Assessment scale (vIGA).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are ≥2 years of age on the day of providing documented informed consent/assent.
2. Have a clinical diagnosis of Atopic Dermatitis (AD) according to the criteria of Hanifin and Rajka (1980) at the Screening visit and a history of AD for at least 6 months (3 months for children under the age of 6).
3. Mild to moderate AD indicated by vIGA (Validated Investigator's Global Assessment) score of 2 (mild) or 3 (moderate) at Screening and at Day 1 prior to application of study intervention.
4. Have AD on the head (including face, but excluding hair-bearing scalp), neck, trunk (excluding groin and genitals), or limbs, covering at least ≥2% of total BSA (body surface area) and not more than 20% at Screening and at Day 1 (Visit 1).
5. Participants who have at least 1 lesion that measures approximately 5 cm2 or more at Screening and Day 1. Lesion must be representative of the participant's atopic dermatitis and not be located on the hands, feet, or genitalia.
6. Have an Eczema Area and Severity Index (EASI) total score of ≥3 to ≤21 at Screening and at Day 1.
7. Have a peak pruritus Numeric Rating Scale (NRS) score of at least 4 at Screening and at Day 1.
8. All allowed oral and topical medications (Protocol Section 6.5) must be stable regimens within the 14 days prior to Day 1.
9. Willing to refrain from using any topical products, including cosmetics and skin cleansers on the AD lesions during the study intervention application period (Section 6.5.1).
10. Participants who are willing and able to comply with all study procedures, including scheduled visits, proper administration of study intervention application, lifestyle considerations.
11. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) OR
    * A WOCBP who agrees to follow the contraceptive guidance in Section 10.4. Male participants are eligible to participate if they agree to follow the contraceptive guidance

Exclusion Criteria:

1. Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to Day 1.
2. Concurrent conditions and history of other diseases:

   1. Any other concomitant skin disorder, pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
   2. The presence of AD lesions only on the hands or feet without prior history of involvement of other classical areas of involvement such as the face or the folds.
   3. Other types of atopic dermatitis.
3. Has recent or anticipated concomitant use of systemic or topical therapies that might alter the course of AD in the opinion of the investigator
4. Ultraviolet (UV) light therapy or prolonged exposure to artificial sources of UV radiation within 2 weeks prior to Screening and/or intention to have such exposure during the study.
5. Use of any of the following treatments within the indicated washout period before Day

   1. 5 half-lives or 12 weeks, whichever is longer - biologic agents (e.g. dupilumab).
   2. 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporin, methotrexate, azathioprine, or other systemic immunosuppressive or immunomodulating agents (e.g. mycophenolate or tacrolimus).
   3. Two weeks - systemic antibiotics.
   4. One week - use of other topical treatments for AD (other than bland emollients).
   5. One week - topical antiviral agents, topical antibacterial agents, topical antifungal agents, topical corticosteroid agents.
   6. One week - oral antibiotics
6. Has undergone treatment within 5 years for any cancer except non-melanoma skin cancers, squamous cell carcinoma, basal cell carcinoma. Participants with adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ are allowed.
7. Active or potentially recurrent dermatologic condition other than AD that may confound evaluation in the opinion of the investigator.
8. Current or recent history (within 3 months) of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease.
9. Have had a systemic infection within the past 3 months requiring hospitalization.
10. Have required the use of parenteral antimicrobial, antivirals, antiprotozoals, antifungals, janus kinase inhibitors (JAK), tyrosine kinase inhibitors (TYK2, or phosphodiesterase 4 (PDE4) inhibitors, monoclonal antibodies (mABs), or other parenteral therapies as judged to be clinically significant by the Investigator within the past 3 months.
11. Has undergone significant trauma or major surgery within 3 months prior to screening or has major surgery planned during the study.
12. Known hypersensitivity to zabalafin or any component of the hydrogel vehicle.
13. Has a presence of depression per the Depression and Anxiety Disorder Score (DASS) scale that is not controlled with medication or is in remission, or the presence of severe depression or suicidal ideation or behavior. Participants with severe depression/suicidal ideation/behavior should be referred to appropriate medical professionals for evaluation.
14. A WOCBP who has a positive serum pregnancy test within 24 hours prior to randomization or treatment allocation.

    Note: If 24 hours have elapsed between the screening pregnancy test and the first dose of study intervention, another serum pregnancy test must be performed and must be negative for participant to start receiving study intervention.
15. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccine and mRNA vaccines are allowed.

    Note: Any licensed COVID-19 vaccine (including for Emergency Use) is allowed in the study if they are Messenger Ribonucleic Acid (mRNA) vaccines, replication-incompetent adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy. Investigational vaccines (ie, those not licensed or approved for Emergency Use) are not allowed.

    Prior/Concurrent Clinical Study Experience:
16. Current treatment or treatment within 90 days or 5 half-lives (whichever is longer) before Day 1 with another investigational medication or current enrollment in another investigational drug protocol.

    Other Exclusion Criteria:
17. Investigator site staff members directly involved in the conduct of the study and their family members; site staff members otherwise supervised by the investigator, are not eligible.
18. Has a history of alcohol or substance abuse within 6 months prior to Screening that in the opinion of the investigator will preclude participation in the study.
19. Have any medical or psychiatric condition which, in the opinion of the Investigator or the Sponsor's Medical Monitor, would place the participant at risk, interfere with participation in the study, or interfere with the interpretation of study results.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of zabalafin hydrogel compared with vehicle in treating mild to moderate AD as assessed by vIGA. | 113 days
  Proportion of participants who achieve Validated Investigator's Global Assessment (vIGA) "clear or almost clear" with a 2-grade improvement from baseline at Day 113.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of zabalafin hydrogel versus vehicle. | 113 days
  * Frequency and severity of Adverse Events (AEs)
  * Study intervention discontinuation due to AEs.
To evaluate the efficacy of zabalafin hydrogel compared with vehicle in treating mild to moderate AD as assessed by absolute change in Eczema area and severity index (EASI) score. | 113 days
  Absolute change in EASI score at Days 15, 29, 57, 85, and 113.
To evaluate the efficacy of zabalafin hydrogel compared with vehicle in treating mild to moderate AD as assessed by vIGA, where response is defined as achieving at least a 1-point decrease from baseline in vIGA score. | 113 days
  Proportion of participants achieving at least a 1-point decrease in vIGA score at Days 15, 29, 57, 85, and 113
To evaluate the efficacy of zabalafin hydrogel compared with vehicle in treating mild to moderate AD as assessed by peak pruritus numerical rating score (NRS), where response is defined as achieving at least a 4-point decrease from baseline. | 113 days
  Proportion of participants achieving at least a ≥4-point decrease in peak pruritus NRS at Days 15, 29, 57, 85, and 113.
To evaluate the efficacy of zabalafin hydrogel compared with vehicle as assessed by Patient oriented eczema measure (POEM) Score, where response is defined as achieving at least a 6-point decrease from baseline. | 113 days
  Proportion of participants achieving at least a ≥6-point decrease in POEM at Days 15, 29, 57, 85, and 113.
To evaluate the antibacterial efficacy of zabalafin hydrogel compared with vehicle in treating mild to moderate AD (Cohort 2). | 113 days
  * Clinical assessment of infection at Days 4, 15, 29, 57, 85, and 113.
  * Bacteriologic assessment of infection at Days 4, 15, 29, 57, 85, and 113.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Pekoe, PhD, Study Director — Alphyn Biologics
Locations (12):
- Australia (12):
  - Canopy Clinical Northern Beaches, Brookvale, New South Wales
  - Momentum Clinical Research, Darlinghurst, New South Wales
  - Premier Specialists, Kogarah, New South Wales
  - St George Dermatology, Kogarah, New South Wales
  - Novatrials, Kotara, New South Wales
  - Innovate Clinical Research, Waitara, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - The Skin Center, Benowa, Queensland
  - Momentum Clinical Research, Wellers Hill, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Canopy Clinical Altona North, North Altona, Victoria
  - Captain Stirling Medical Centre, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alphyn announces positive results from second cohort of phase 2a clinical trial in atopic dermatitis. News release. PR Newswire. March 7, 2024. — https://www.prnewswire.com/news-releases/alphyn-announces-positive-results-from-second-cohort-of-phase-2a-clinical-trial-in-atopic-dermatitis-302082303.html
- See also: Alphyn Granted U.S. Patent Covering First-in-Class Treatment for Atopic Dermatitis — https://alphynbiologics.com/press-release/alphyn-granted-u-s-patent-covering-first-in-class-treatment-for-atopic-dermatitis/